CLINICAL TRIAL: NCT02959424
Title: Quality of Life Among Patients With Chronic Esophageal Disorders : Spanish Translation and Validation of the Survey "Northwestern Esophageal Quality of Life Scale" in Hispanics
Brief Title: NEQOL Survey Spanish Validation in a Hispanic Clinic Based Population
Status: Completed | Type: Observational
Sponsor: Carlos Robles-Medranda (Other)
Responsible Party: Sponsor-Investigator, Carlos Robles-Medranda, MD, Instituto Ecuatoriano de Enfermedades Digestivas
Organization: Instituto Ecuatoriano de Enfermedades Digestivas (Other)
Other Study IDs: NOV-7-2016
Record Dates: First submitted 2016-11-07; First posted 2016-11-09 (Estimated); Last update posted 2018-08-09 (Actual); Status verified 2018-08

CONDITIONS: Gastroesophageal Reflux Disease and Esophageal Motility Disorders
MeSH Terms: conditions — Gastroesophageal Reflux; Esophageal Motility Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Spanish Northwestern Esophageal Quality of Life questionnaire
  Other Names: Spanish NEQOL

SUMMARY:
Chronic esophageal disorders affect approximately one third part of global population, with a deleterious impact in the quality of life of patients. Measured of health related quality of life in chronic esophageal conditions such as gastroesophageal reflux disease and achalasia are widely used to measure this important patient-reported outcome. The Northwestern Esophageal Quality of Life (NEQOL) is a hybrid measure of esophageal illness, allowing for broad use across esophageal diseases while maintain sensitivity to nuances of a specific condition. The NEQOL is a reliable and valid hybrid measure of disease specific health related quality of life across several chronic esophageal conditions. The Ecuadorian Institute of Digestive Diseases aims to translate and validate this survey into Spanish for its use in a Hispanic population. This cross-sectional study aims to translate, apply and validate the NEQOL in the patients attending in the esophageal division of the institute.

DETAILED DESCRIPTION:
Methods: An authorization for translating the survey into Spanish was obtained from the survey authors. The translation and cross-cultural adaptations were carried out based on guidelines and international criteria proposed by Sperber. The NEQOL was translated independently from English into Spanish by two professional translators. Each one provided a written report, which was combined by the authors in a new version that contained the most reliable translation for each question. The new version was back translated to English by two different professional translators, who were blinded to the original version of the NEQOL. A new English version was developed by combining the written reports. The aim of the back translation was to compare each item of the new English version with the original NEQOL. Each item of the new English version was compared with the original questionnaire by 30 native English speakers. The success of the translation was evaluated using two scales of comparison: comparability of language and similarity of interpretability. Each one used Likert scales ranging from 1 (extremely comparable/ extremely similar) to 7 (not at all comparable/ not at all similar). A mean score for each question was obtained. Questions with mean scores of three or less were included in the Spanish version. The Spanish version of the NEQOL was tested on 10 subjects diagnosed with GERD, each subject provided feedback on the survey content, which was used to make final corrections. The questionnaire contains fourteen questions; every statement refers to the impact of the esophageal condition in the quality of life. There are five options ranking from not at all true to very true, with every option meaning a numerical value, a higher grade in the questionnaire will express a better quality of life and a low impact in the health-related quality of life.

Patients above 18 years old with chronic esophageal disorders, that require a functional esophageal test such as ph-impedanciometry and/or high-resolution manometry, will be included. Written informed consent will be obtained. All participants will complete the questionnaire before performing the functional esophageal tests and a gastroenterologist specialized on functional esophageal pathology will perform the esophageal tests and analyze the results. Finally, the data from the questionnaire will be compared with the esophageal tests results in order to stablish if there is a correlation between the impact in the quality of life measured by the questionnaire and the tests results.

Statistical analysis: Base line characteristics will be analyzed using Chi-square o Fisher Test for categorical variable, and the Mann-Whitney Test for continuing variables. Continuous variables will be expressed as mean +/- standard deviation. The sensitivity, specificity, predictive values and accuracy will be calculated with the 95% Confidence Interval (95% CI). A P value of less than 0.05 was considered to be statistically significant. All the statistical analysis was performed using SPSS software suite v.22.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent obtained
* Ability to complete the survey
* Hispanic patients above 18 years old with chronic esophageal disorders, that require a functional esophageal test such as ph-impedanciometry and/or high-resolution manometry

Exclusion Criteria:

* Not able to complete the survey
* Not in the range of age acceptable for inclusion

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hispanic patients above 18 years old with chronic esophageal disorders, that require a functional esophageal test such as ph-impedanciometry and/or high-resolution manometry
Sampling Method: Non-Probability Sample
Enrollment: 385 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-10 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
To measure the disease related quality of life and its impact among patients with chronic esophageal disorders by translating and validating into Spanish the Northwestern Esophageal Quality of Life Scale survey. | 9 month

CONTACTS AND LOCATIONS:
Overall Officials: Carlos A Robles-Medranda, MD, Principal Investigator — Ecuadorian Institute of Digestive Diseases
Locations (1):
- Ecuadorian Institute of Digestive Diseases, Omnihospital, Guayaquil, Guayas, Ecuador

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] El-Serag HB, Sweet S, Winchester CC, Dent J. Update on the epidemiology of gastro-oesophageal reflux disease: a systematic review. Gut. 2014 Jun;63(6):871-80. doi: 10.1136/gutjnl-2012-304269. Epub 2013 Jul 13. PMID 23853213
- [Result] O'Neill OM, Johnston BT, Coleman HG. Achalasia: a review of clinical diagnosis, epidemiology, treatment and outcomes. World J Gastroenterol. 2013 Sep 21;19(35):5806-12. doi: 10.3748/wjg.v19.i35.5806. PMID 24124325
- [Result] Bedell A, Taft TH, Keefer L, Pandolfino J. Development of the Northwestern Esophageal Quality of Life Scale: A Hybrid Measure for Use Across Esophageal Conditions. Am J Gastroenterol. 2016 Apr;111(4):493-9. doi: 10.1038/ajg.2016.20. Epub 2016 Feb 16. PMID 26881974
- [Result] Roman S, Gyawali CP, Xiao Y, Pandolfino JE, Kahrilas PJ. The Chicago classification of motility disorders: an update. Gastrointest Endosc Clin N Am. 2014 Oct;24(4):545-61. doi: 10.1016/j.giec.2014.07.001. Epub 2014 Aug 1. PMID 25216902